CLINICAL TRIAL: NCT02614079
Title: Evaluation of the Percutaneous Spinal Cord Stimulation Trial Using the Dermatomal Somatosensory Evoked Potentials (DSSEP) Collision Testing
Brief Title: Evaluation of the Percutaneous SCS Trial Using the DSSEP Collision Testing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment. Futility.
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Atallah SCS DSSEP
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-01

CONDITIONS: Back Pain With Radiation
Keywords: lumbago; low back pain; leg pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- DSSEP (Experimental): DSSEP testing after SCS trial lead placement
  Interventions: Device: DSSEP

INTERVENTIONS:
Device: DSSEP — Collision testing after the placement of SCS leads

SUMMARY:
This study is to objectively evaluate the success of a spinal cord stimulator (SCS) trial using testing (DSSEP) to determine if the paresthesia (tingling sensation) or pain reduction achieved correlates with the degree of stimulation.

DETAILED DESCRIPTION:
The SCS trial leads will be placed as per standard of care, using fluoroscopic guidance and leads will be checked for proper positioning. Leads will be tested for appropriate paresthesia coverage of the patient's painful area(s), using multiple electrode configurations and lead positions (dependent on the location of the pain). After the leads are secured, the patient will be sent to the recovery room where the DSSEP test will be performed. A technologist will glue/tape recording electrodes to the patient's head, neck, back or legs. One or two stimulating electrodes are also placed on the patient's leg. Each electrode is checked with a meter to ensure proper functioning. Pulsing stimulus will start in one of the stimulating electrodes. Each time a different area is tested, the pulsing will be started again. Each area tested will take 10-15 minutes. The painful dermatomal distribution area, specific to each patient will be used for dermatomal SSEP stimulation. Placement will be correlated with nerve roots involved with the corresponding dermatomes. Measurements will be obtained to determine collision criteria.

ELIGIBILITY:
Inclusion Criteria

A subject will be eligible for inclusion in this study only if all the following criteria apply:

A. Subject understands the procedures, agrees to participate in the study, and has signed and dated the informed consent form prior to the initiation of any study-related activities.

B. Subjects are male or female greater than 18 years old at the time of screening visit.

C. Pain in one or both lower extremities. D. Pain is not responding to conservative treatment such as physical therapy or medications.

E. Average pain rating of at least 4 on a scale 0 to 10, on average, prior to enrollment in the study.

F. Patient is mentally competent to make decisions.

Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

A. Female subject with childbearing potential (a premenopausal female, who is not surgically sterile).

B. Subjects who poorly cooperate or have any cognitive impairment. C. Patient with severe concomitant depression. D. Inability to communicate adequately with physician and /or study coordinator.

E. Patient is diagnosed with a psychiatric condition that will likely interfere with diagnostic accuracy of the workup protocol or with recovery following the anticipated procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph N Atallah, MD, Principal Investigator — Universtiy of Toledo
Locations (1):
- University of Toledo, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The study was terminated early due to lack of enrollment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from subjects scheduled to receive the Spinal Cord stimulator (SCS) trial leads at the University of Toledo Medical Center.
Pre-assignment Details: 6 participants were enrolled.
Groups:
- DSSEP - Dermatomal Somato Sensory Evoked Potentials: DSSEP testing after SCS trial lead placement
  DSSEP: Collision testing after the placement of SCS leads
Period: Overall Study
Arm/Group | DSSEP - Dermatomal Somato Sensory Evoked Potentials
Started | 6
Completed | 5 (1 participant withdrew from the study prior to completion of DSSEP testing)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | DSSEP
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Collision
Description: Positive collision: 75% or greater decrease in amplitude from the baseline waveform. Centroparietal (CPz)-Popliteal Fossa (Fpz) cortical montage (images) will be used as primary montage to evaluate collision results.
Time Frame: Day 1
Population: 5 participants completed DSSEP testing after placement of SCS Trial leads.
Measure: Count of Participants; unit: Participants
Arm/Group | DSSEP
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 4 hours after DSSEP testing performed. All cause mortality not monitored/assessed.
Description: No adverse events reported. All cause mortality not monitored/assessed.
Arm/Group | DSSEP
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes